CLINICAL TRIAL: NCT03354091
Title: Active@Work - Optimizing Physical Activity at Work With Personalized Decision Support Among Individuals With Osteoarthritis.
Brief Title: Active@Work - Optimizing Physical Activity at Work.
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Lund University (Other)
Collaborators: Halmstad University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 2016-02327
Record Dates: First submitted 2017-11-15; First posted 2017-11-27 (Actual); Last update posted 2021-03-04 (Actual); Status verified 2021-03

CONDITIONS: Osteoarthritis, Knee; Osteoarthritis, Hip; Physical Activity
MeSH Terms: conditions — Osteoarthritis, Knee; Osteoarthritis, Hip; Motor Activity

STUDY DESIGN:
Intervention Model Description: Cluster-Randomized controlled trial
Who Masked: Investigator
Masking Description: Masking is performed through sealed envelopes. The investigator has no knowledge of which patients who is randomized to intervention or control
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention (Experimental): Patient education program and the use of an Fitbit where the users can monitore their activity and receive minor feedback regarding physical activity.
  Interventions: Device: FitBit Flex 2
- Control (No Intervention): Patient education program only.

INTERVENTIONS:
Device: FitBit Flex 2 — Participants in the intervention Group will wear the FitBit Flex 2 for Three months.
  Arms: Intervention

SUMMARY:
The aim of this project is to explore if monitoring physical activity including feedback can have any effect on physical activity level, function, work ability, health related quality of life or work productivity among individuals with hip and/or knee osteoarthritis. This will be performed by evaluating the use of mobile technology and activity monitoring to support physical activity in individuals with OA in a cluster randomized controlled trial. The investigators research questions are:

• Can an intervention, comprised of the above mentioned technology, have any effect on physical activity level, function, work ability, quality of life or work productivity among individuals with OA?

DETAILED DESCRIPTION:
Methods Design and setting The project will be performed as a cluster randomized controlled intervention study within primary health care in the region of Skåne and Halland.

Sample Patients who are referred to the patient education program for OA in primary health care will be invited to participate in the project. Participants will also be recruited using advertisement on social media. Participants recruited from social media will attend the patient education program for OA arranged by this project.

There will be one control group and one intervention group, see details below:

A. Patient education program and physical activity monitoring. C. Patient education program (control).

Each group within the patient education program for OA will be randomized to either group A or group C. Patients that fulfil the inclusion criteria will then be asked to participate. Digital (BankID or e-legitimation) informed consent will be obtained at the project's website. Recruitment of participants in intervention group A and control group C starts in autumn 2017 and continues through spring 2019 or when sufficient numbers of participants have been included.

Interventions Activity monitoring will be performed by giving each participant in group (A) a wearable sensor (Fitbit Flex 2), where the daily physical activity level will be recorded. The monitoring will start at the patient education program within BOA. All activity monitors will be programmed with a daily goal of 7 000 steps. The participants will have the opportunity to follow their physical activity through the fitbit app were they also will receive standardised feedback. The intervention will be performed during three months, with follow-ups online after 3, 6 and 12 months.

Measures Patient-reported outcomes

Participants will answer the following questionnaires at baseline, after the intervention (3 months) and 6 and 12 months after baseline. Measurements will include:

* Self-rated work ability (Work ability Index, Ilmarinen,2007)
* Self-rated work productivity (WPAI-OA, Legget et.al.,2016)
* Self-rated health-related quality of life (EQ-5D) (http://www.euroqol.org/)
* Self-rated function in relation to hip and knee arthrosis (HOOS, Nilsdotter 2003, KOOS, Paradowski 2006).
* Self-rated physical activity (IPAQ, Craig et.al.2003).
* Questions about the work environment and physical activity.

Statistics The investigators will recruit approximately 80 participants/group. With this sample size and 80 % power, effect sizes of about 0.45 SD (significance level 5%) can be identified. In terms of WAI, this corresponds to SD 6, approximately 2,7 points increase/higher score in the intervention group, compared to the control group. Compliance with the intervention will comprise of the activity monitoring device used on at least 50% of the work days. With relatively large group sizes and most data expected to a follow an approximately normal distribution, group differences in the development over time with respect to the different outcome variables will be analyzed by ANOVA models (repeated measures or cross sectional comparison of mean difference scores). Some outcome variables, may likely be skewed and hence appropriate transformations, or non-parametric models, will be applied. Final and exact analytical strategies will be decided once data is available for exploration of final group sizes and distributions/symmetry of numeric outcome variable data.

ELIGIBILITY:
Inclusion Criteria:

* Working at least 50 %

Exclusion Criteria:

* Not being able to do physical activity, non-Swedish speaking

Ages: 18 Years to 67 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 160 (Actual)
Dates: Start 2017-11-16 (Actual); Primary Completion 2020-05-30 (Actual); Study Completion 2020-06-15 (Actual)

PRIMARY OUTCOMES:
Change in work ability | Baseline, 3 months, 6 months, 12 months
  Questionnaire Work ability index (WAI) 7-49 points. 7-27 points (bad) - restore work ability. 28-36 points (moderate) - improve work ability. 37-43 points (good) - support work ability. 44-49 points (very good) - support work ability.

SECONDARY OUTCOMES:
Change in physical activity | Baseline, 3 months, 6 months, 12 months
  Questionnaire: International physical activity questionnaire (IPAQ). Three levels of physical activity; Category 1: Low. This is the lowest level of physical activity. Those individuals who not meet criteria for categories 2 or 3 are considered low/inactive.
  Category 2: Moderate. Any one of the following 3 criteria:
  * 3 or more days of vigorous activity of at least 20 minutes per day OR
  * 5 or more days of moderate-intensity activity or walking of at least 30 minutes per day OR
  * 5 or more days of any combination of walking, moderate-intensity or vigorous intensity activities achieving a minimum of at least 600 MET-min/week.
  Category 3: High. Any one of the following 2 criteria:
  * Vigorous-intensity activity on at least 3 days and accumulating at least 1500 MET-minutes/ week OR
  * 7 or more days of any combination of walking, moderate-intensity or vigorous intensity activities achieving a minimum of at least 3000 MET-minutes/week
Change in work productivity | Baseline, 3 months, 6 months, 12 months
  Questionnaire: Work Productivity and Activity Impairment Questionnaire - osteoarthritis (WPAI - OA) WPAI outcomes are expressed as impairment percentages, with higher numbers indicating greater impairment and less productivity, i.e., worse outcomes, as follows: Questions:
  1. = currently employed
  2. a = hours missed due to specified problem
  2b = hours missed due to other health problems 2c = hours missed other reasons 3 = hours actually worked 4a = degree problem affected productivity while working 4b = degree other health problems affected productivity while working 5a = degree problem affected regular activities 5b = degree other health problems affected regular activities
  Scores:
  Multiply scores by 100 to express in percentages.
Change in quality of life | Baseline, 3 months, 6 months, 12 months
  Questionnaire EQ5D. EuroQol. The EQ5D consists of a scale from 0-100 where 0 is the worst Health and 100 is the best. There is also an additional five questions from where a Health-index is calculated with a mathematic formula. The Health-index ranges from 1 to -0,594. 1 is best.
Change in function of Hip or knee | Baseline, 3 months, 6 months, 12 months
  Questionnaire: Hip/Knee disability and Osteoarthritis Outcome Score (HOOS/KOOS). A total sum of 100 indicate no problems and 0 indicate extreme problems.

CONTACTS AND LOCATIONS:
Overall Officials: Frida Eek, Ass prof, Principal Investigator — Lund University
Locations (1):
- Vårdcentralen Dalby, Dalby, Sweden

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Ostlind E, Eek F, Stigmar K, Ekvall Hansson E. Effects of self-monitoring physical activity with wearable activity trackers on perceived joint function and health-related quality of life in people with hip and knee osteoarthritis: a secondary analysis of a cluster-randomised clinical trial. BMC Musculoskelet Disord. 2025 Jan 9;26(1):33. doi: 10.1186/s12891-024-08238-8. PMID 39789623
- [Derived] Ostlind E, Eek F, Stigmar K, Sant'Anna A, Hansson EE. Promoting work ability with a wearable activity tracker in working age individuals with hip and/or knee osteoarthritis: a randomized controlled trial. BMC Musculoskelet Disord. 2022 Feb 3;23(1):112. doi: 10.1186/s12891-022-05041-1. PMID 35114983